CLINICAL TRIAL: NCT04506268
Title: Opt-In Versus Opt-Out for COVID Screening Assessment for Exposure
Brief Title: COVID-19 SAFE Enrollment
Acronym: COVID SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 843565
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID-19; Coronavirus; opt-in; opt-out; behavioral science
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opt-in Recruitment Email (Experimental): Participants will receive a recruitment email that describes the objectives of a new COVID-19 voluntary screening program, and invites them to enroll.
  Interventions: Behavioral: Opt-in Recruitment Email
- Opt-out Recruitment Email (Experimental): Participants will receive a recruitment email that describes the objectives of a new COVID-19 voluntary screening program, and informs them that they have been conditionally enrolled.
  Interventions: Behavioral: Opt-out Recruitment Email

INTERVENTIONS:
Behavioral: Opt-out Recruitment Email — Behaviorally informed, opt-out framed recruitment email
  Arms: Opt-out Recruitment Email
Behavioral: Opt-in Recruitment Email — Standard, opt-in framed recruitment email
  Arms: Opt-in Recruitment Email

SUMMARY:
In order to safely and effectively reopen businesses and universities across the US, institutions will need to develop approaches to rapidly identify COVID-19 cases and manage their spread while balancing program effectiveness, feasibility, costs, and scalability.

The investigators will evaluate the implementation of a COVID-19 screening program that coordinates several existing systems at the University of Pennsylvania including saliva-based viral testing and test different outreach strategies (opt-in vs opt-out) to improve program enrollment.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has resulted in close to 10,000,000 reported cases worldwide, including more than 2,000,000 aggregated reported cases and 120,000 deaths in the United States. Initial efforts to address the COVID-19 pandemic were aimed at testing symptomatic individuals, implementing stay-in-place orders, and at increasing hospital capacity to meet surge demands. While the US continues to confront the current crisis, we must plan for the future by putting in place tools to enhance our ability to conduct effective screening, containment, and case management.

Widespread COVID-19 testing is needed to safely and effectively reopen schools and businesses across the US. However, currently approved testing options require reagents that are limited in supply, severely hindering scalability. Emerging evidence indicates that saliva testing with the option of at-home sample collection can accurately identify COVID-19 viral infection. Additional diagnostic testing options will continue to increase patient access. Moreover, this approach provides an option for the easy, safe and convenient collection of samples required for testing without traveling to a doctor's office, hospital, or testing site. Collection by the patient also reduces exposure of health care workers to the virus and preserves limited personal protective equipment.

With access to expanded testing, health systems and universities will need to test alternative methods to manage COVID-19 spread while balancing program effectiveness, feasibility, costs, and scalability. Insights from the field of behavioral economics offer promise for designing and sustaining these kinds of policies. Specifically, research has demonstrated that an opt-out framed recruitment strategy compared to a conventional opt-in strategy can improve enrollment and adherence to behavioral interventions.

For these reasons, the investigators propose to evaluate the implementation of a COVID-19 screening program that uses saliva-based testing and to test approaches to improve program enrollment.

ELIGIBILITY:
Inclusion Criteria:

•University of Pennsylvania staff, faculty, and trainees that have returned to work on campus who have been identified by leadership at the University of Pennsylvania Perelman School of Medicine.

Exclusion Criteria:

•Participants will not be eligible for the study if they identify any reason they are unable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion Enrolled | 4 weeks
  The proportion of those invited that enroll in the study

SECONDARY OUTCOMES:
Participant Age | 4 weeks
  The average age of participants enrolled in the study
Participant Sex | 4 weeks
  The proportion of females enrolled in the study
Participant Race/Ethnicity | 4 weeks
  The proportion of enrolled participants belonging to specified categories of race (e.g., Alaska Native, Asian, Black or African American, Native Hawaiian or other Pacific Islander, White or Caucasian) and ethnicity (i.e., Hispanic or Latino, Non-Hispanic or Latino)
Participant Income | 4 weeks
  The proportion of enrolled participants belonging to specified categories of income (e.g., Less than $10000, $10000 to $19999, $20000 to $29999, $150000 or more)
Participant Education | 4 weeks
  The proportion of enrolled participants belonging to specified categories of education (e.g., less than high school, some high school, high school grad, college: 4 year degree, post-college education)
Test Completion | 8 weeks
  The proportion of enrolled participants that submit a saliva sample

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S Patel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No